CLINICAL TRIAL: NCT04888117
Title: COMPlex Cholecystectomy Trial (COMPaCT): A Prospective Multi-Center Study of Short-Term Outcomes After Complex Cholecystectomy
Brief Title: Prospective Multi-Center Study of Short-Term Outcomes After Complex Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: COMPaCT
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-01

CONDITIONS: Laparoscopic Cholecystectomy; Robotic-assisted Cholecystectomy
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Laparoscopic cholecystectomy: Subject has a diagnosis of acute cholecystitis and is admitted through the ER for a laparoscopic cholecystectomy.
  Interventions: Procedure: Laparoscopic cholecystectomy
- Robotic-assisted cholecystectomy: Subject has a diagnosis of acute cholecystitis and is admitted through the ER for a robotic-assisted cholecystectomy.
  Interventions: Procedure: Robotic-assisted cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — With the patient under general anesthesia, several small incisions are made in the abdomen. Ports are placed, the abdomen is insufflated, and laparoscopic instruments as well as a laparoscope are inserted to complete the cholecystectomy according to the surgeon's standard practice.
  Groups: Laparoscopic cholecystectomy
Procedure: Robotic-assisted cholecystectomy — With the patient under general anesthesia, several small incisions are made in the abdomen. Ports are placed, the abdomen is insufflated, and the da Vinci Robotic Surgical System (Intuitive) is docked to the patient and used to complete the cholecystectomy according to the surgeon's standard of care.
  Groups: Robotic-assisted cholecystectomy

SUMMARY:
The study aims to evaluate the short-term clinical outcomes after complex robotic-assisted and laparoscopic cholecystectomies.

DETAILED DESCRIPTION:
This is a multi-center cohort study, evaluating short-term clinical outcomes after complex robotic-assisted and laparoscopic cholecystectomies. The primary outcomes include the rate of conversion to open, rate of intra-operative adverse events, the rate of post-operative adverse events relating to the cholecystectomy within 30 days, and re-admissions and re-operations relating to the cholecystectomy within 30 days. In addition, operative time, the rate of use of intra-operative imaging, the hospital length of stay, and pain and QOL scores will be collected as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 and 80 years of age at the time of surgery
2. Subject is a candidate for a cholecystectomy
3. Subject has a diagnosis of acute cholecystitis and is being admitted through the Emergency Room (ER)

Exclusion Criteria:

1. A single port (single site or single incision procedure) cholecystectomy will be performed
2. Subject will undergo a concomitant procedure
3. Subject is contraindicated for surgery or a minimally invasive approach
4. Subject has a known bleeding or clotting disorder that is not able to be controlled during surgery
5. Pregnant or suspect pregnant
6. Subject is mentally handicapped or has a psychological disorder or severe systematic illness that would preclude compliance with the study requirements or ability to provide informed consent
7. Subject belonging to other vulnerable population, e.g. prisoner or ward of the state
8. Subject is unable to comply with the follow-up visit schedule
9. Subject is currently participating in another research study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who are eligible based on the inclusion/exclusion criteria may participate in the study. Approximately 100 subjects will be enrolled in each cohort (laparoscopic and robotic-assisted). In each cohort, a maximum of 50% of subjects may be enrolled with a Nassar Grade II, and a minimum of 50% of subjects with either Nassar Grade III or IV may be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Conversion to open | Intra-operative
  The rate of conversion of the cholecystectomy to open, defined as robotic-assisted surgery converted to an open approach
Number of adverse events | Intra-operative through the 30 days follow-up period
  Intra-operative or post-operative adverse events related to the cholecystectomy
Re-admissions | After discharge from the hospital post-procedure through the 30 days follow-up period
  Re-admissions to the hospital related to the cholecystectomy through the 30 days follow-up period
Re-operations | After the procedure but prior to discharge, through the 30 day follow-up period
  Re-operations related to the cholecystectomy through 30 days follow-up

SECONDARY OUTCOMES:
Operative time | Intra-operative
  Operative time, defined as first incision to closure of the incision
Use of intra-operative imaging | Intra-operative
  The rate of intra-operative imaging, including indocyanine green fluorescent imaging and cholangiography
Length of hospital stay | From admission to discharge, up to approximately one week
  How long the patient was admitted to the hospital
Biliary anatomy identification | Intra-operative
  Ability for surgeons to identify biliary anatomy and incidence of abnormal biliary anatomy intra-operatively
Change in pain score assessed by the PROMIS 3a from baseline to 14 days | 14 days
  Change in patient reported pain scores assessed by the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a survey, with a scale from 1-5; 1 meaning no pain and 5 meaning severe pain
Change in pain score assessed by the PROMIS 3a from baseline to 30 days | 30 days
  Change in patient reported pain scores assessed by the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a survey, with a scale from 1-5; 1 meaning no pain and 5 meaning severe pain
Change in Quality of Life assessment: EQ-5D-5L (EQ) from baseline to 14 days | 14 days
  Quality of life using the EQ-5D-5L (EQ) assessment tool, with scores on individual questions ranging from no problems to extreme problems, with a scale of health ranging from 0 (the worst health you can imagine) to 100 (the best health you can imagine)
Change in Quality of Life assessment: EQ-5D-5L (EQ) from baseline to 30 days | 30 days
  Quality of life using the EQ-5D-5L (EQ) assessment tool, with scores on individual questions ranging from no problems to extreme problems, with a scale of health ranging from 0 (the worst health you can imagine) to 100 (the best health you can imagine)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Baptist Health-South Florida, Miami, Florida
  - Progressive Surgical Associates, Silver Cross Hospital, New Lenox, Illinois
  - Lovelace Medical Group, Albuquerque, New Mexico
  - St. David's Healthcare, Austin, Texas